CLINICAL TRIAL: NCT05971927
Title: The Effect of Simulation Teaching Method on Vaginal Examination Practice Skills and Self-Confidence Development in Labor in Midwifery Students
Brief Title: Simulation Teaching Method and Vaginal Examination in Midwifery Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Döndü BATKIN ERTÜRK, doctoral lecturer, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: TOKAT02
Record Dates: First submitted 2023-07-17; First posted 2023-08-02 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Vaginal Examination
Keywords: Midwifery student; Vaginal examination; Confidence; Skill; Simulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Simulation education
  Interventions: Behavioral: Simulation education
- Control groups (No Intervention): The control group did not receive any simulation training.

INTERVENTIONS:
Behavioral: Simulation education — Randomly assigned experimental group students performed eight different vaginal examination scenarios in the laboratory on the fetal monitoring and labor progress model set for cervical dilatation, cervical effacement, presenting fetal part, presence of amniotic membrane and fetal descent. The researchers repeated the vaginal examination scenario and informed the students about the evaluation results after each student had performed the vaginal examination scenario prepared by the researchers. This process continued until the experimental group students completed eight different vaginal examination scenarios.
  Arms: Experimental group

SUMMARY:
This study was planned to evaluate the effect of simulation teaching method on the ability to apply vaginal examination in labor and self-confidence in midwifery students.

DETAILED DESCRIPTION:
Two skills, abdominal palpation and vaginal examination, are used to clinically monitor the progress of labor. Vaginal examination is the most accepted method to measure the progress of labor.Vaginal examination, which is routinely applied in the evaluation of labor progress, is an important part of midwifery care. However, it is reported that the accuracy level of vaginal examination for new students is low. This essential skill is a learned tactile/tactile skill that requires consistency to properly manage women in labor. Therefore, it cannot be learned through observation alone; In order to acquire this skill, students need to perform a large number of vaginal examinations in women who have given birth. The usual/classic training technique for teaching vaginal examination is that the midwifery student performs a vaginal examination on the woman in labor under the supervision of an experienced obstetrician, and then the experienced obstetrician repeats this examination to determine the accuracy of the trainee student's assessment. Simulation-based learning improves the understanding, retention and active use of knowledge and skills, reduces the student's pre-application anxiety, and increases self-confidence. It is seen that simulation, which has been widely used in medical education in recent years, is also used as a teaching method in the development of practice skills of midwifery students.There are several studies in the literature evaluating the effect of simulation training on students' vaginal examination skills and self-confidence.In a study conducted to evaluate the benefits of simulation training in teaching obstetric vaginal examination techniques to medical students, it was found that the vaginal examination accuracy of students who received simulation training was significantly higher than those who did not receive simulation training. In this study, it was concluded that simulation training helped inexperienced students improve their vaginal examination skills before performing such procedures on real patients, interns who performed simulated examination showed significantly higher accuracy in vaginal examination evaluations than the control group. However, according to the available data, no study has been found that examines the effect of simulation training on vaginal examination skills in midwifery students.

This study was planned to evaluate the effect of simulation teaching method on the ability to apply vaginal examination in labor and self-confidence in midwifery students.

Type of Study: The study was planned as a randomized controlled trial.

Place and Time of the Research: The research was carried out at Tokat Gaziosmanpaşa University Faculty of Health Sciences, Tokat Gaziosmanpaşa University Health Research and Application Hospital and Tokat Provincial Health Directorate Tokat State Hospital between 10.02.2020-17.05.2020.

Population and Sample of the Research:

The universe of the research consisted of 66 students who took the Normal Birth and Postpartum Period and Risky Birth and Postpartum Period course for the first time in the Department of Midwifery, Faculty of Health Sciences, Tokat Gaziosmanpaşa University.

Students who agreed to participate in the study voluntarily were included in the study.

66 midwifery students forming the research sample were ranked from high to low according to their general academic grade point average. After the group with the highest grade point average was determined randomly (by drawing lots), the students were assigned to the experimental and control groups, respectively.

Data Collection Tools

The Effect of Simulation Teaching Method on Vaginal Examination Practice Skills and Self-Confidence Development in Midwifery Students Questionnaire The questionnaire consists of three parts.

A. Socio-demographic characteristics of students

In this section, midwifery students' age, marital status, graduated school, family structure, place of residence, education level of the mother and father, perception of income, where the family lives, the presence of health personnel in the family members, their position, if any, their satisfaction with the midwifery department. There are a total of 18 questions about how they evaluate the difference between the preference order of the midwifery profession, the general academic grade point average, the level of finding sufficient theoretical knowledge and skills in vaginal examination, previous vaginal examination practice and examination findings, and the findings of an experienced obstetrician.

B. Students' self-confidence ratings on performing the vaginal examination application steps This is the section in which the students rank their self-confidence in performing the vaginal examination application steps (22 items) prepared by the researchers by examining the literature. It is scored as I do not trust myself at all-1, I do not trust myself-2, I have little confidence in myself-3, I have confidence in myself-4, I am very confident in myself-5.C. Vaginal examination evaluation results of the students in the clinic

C. Vaginal examination evaluation results of the students in the clinic This is the section where the evaluation results (cervical effacement, cervical dilatation, presence of amniotic membrane, presenting fetus part and fetal descent) of the midwifery student and experienced health professional (midwife, nurse and doctor) in vaginal examinations performed on women in the clinic for both groups are recorded.

Application of the Research:

All students who took the Normal Birth and Postpartum Period and Risky Birth and Birth and Postpartum Period courses were given a theoretical lecture on the steps of vaginal examination in labor and the criteria to be evaluated in vaginal examination, and a video on the subject was watched.

After giving information about the study, informed consent was obtained from all students who voluntarily agreed to participate in the study.

The students were asked to fill in the questionnaires prepared by the researchers, examining the socio-demographic characteristics and vaginal examination experiences of the students, and to rate their self-confidence in performing the vaginal examination application steps.

The experimental group students, which were determined as random, performed eight different vaginal examination scenarios on the fetal monitoring and labor progress model set in terms of cervical effacement, dilatation and the presence of the presenting part and amniotic sac.

The control group did not receive any simulation training.

The students in both groups were asked to rate their self-confidence in performing the steps of performing the vaginal examination for the second time before performing the first vaginal examination on the woman in the clinic.

Vaginal examination results (cervical effacement, cervical dilatation, presence of amniotic membrane, presenting fetus part, and fetal descent) of the midwifery student and experienced health professional (midwife, nurse and doctor) were recorded in the vaginal examinations performed on women in the clinic for both groups.

In this study, the vaginal examination procedure normally used by midwifery students during their professional practice in health institutions was used.

An experienced health professional performed the vaginal examination in the woman in labor, then the midwifery student repeated the vaginal examination on the same woman under the supervision of an experienced health professional and the evaluation findings were compared.

Informed consent was obtained from the women before the vaginal examination, infection control measures were taken during the examinations (hand washing, wearing sterile gloves and avoiding frequent vaginal examinations), and the privacy of the women was respected as much as possible. The findings of experienced health professionals were accepted as the gold standard in the study. Student findings consistent with the findings of the experienced healthcare professional were evaluated as correct, and student findings that were not compatible with or could not be evaluated with the findings of the experienced healthcare professional were evaluated as incorrect.

Evaluation of Research Data:

Descriptive statistics were calculated to give information about the general characteristics of the research groups. Qualitative data were expressed as percentages and compared using the Chi-Square Test or the Fisher Exact Test. Quantitative data were expressed as mean±standard deviation, and were compared using the Independent Two-Group T-Test. P<0.05 was considered statistically significant. Calculations were made with ready-made statistical software.

Ethical Aspect of Research:

Institutional permission from Tokat Gaziosmanpaşa University Faculty of Health Sciences, Tokat Gaziosmanpaşa University Health Research and Application Hospital and Tokat Provincial Health Directorate Tokat State Hospital and Tokat Gaziosmanpaşa University Clinical Research Ethics Committee approval were obtained for the research. Informed consent was obtained from all participants (midwifery students and women in labor) who would participate in the study.

Parameters Students' self-confidence ratings in performing the vaginal examination application steps

-Vaginal examination evaluation parameters (cervical effacement, cervical dilatation, presence of amniotic membrane, presenting fetus part and fetal descent)

ELIGIBILITY:
Inclusion Criteria:

* Midwifery students enrolled in Normal Birth and Postpartum Term Course in the 2019-2020 academic year

Exclusion Criteria:

* Students who did not volunteer to participate in the study
* Students who did not perform vaginal examination on real women at the clinic

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Students' self-confidence ratings in performing the vaginal examination application steps | At the beginning of the study
  I am not at all confident-1 I am not confident-2 I have little confidence in myself-3 I am confident-4 I am very confident-5 In the analysis of students' self-confidence in performing the vaginal examination practice steps, the categories of "I am not at all confident", "I am not confident" and "I have little confidence in myself" were combined as "low self-confidence", while the categories of "I am confident" and "I am very confident" were combined as "high self-confidence".
  Each step was evaluated separately.
Students' self-confidence ratings in performing the vaginal examination application steps | Within 1-6 months after the start of the study
  I am not at all confident-1 I am not confident-2 I have little confidence in myself-3 I am confident-4 I am very confident-5 In the analysis of students' self-confidence in performing the vaginal examination practice steps, the categories of "I am not at all confident", "I am not confident" and "I have little confidence in myself" were combined as "low self-confidence", while the categories of "I am confident" and "I am very confident" were combined as "high self-confidence".
  Each step was evaluated separately.
Cervical effacement | Within 1-6 months after the start of the study
  as a percentage (accurate and wrong)
Cervical dilatation | Within 1-6 months after the start of the study
  in centimeters (accurate and wrong)
Presenting fetal part | Within 1-6 months after the start of the study
  head, breech etc. (accurate and wrong)
Presence of amniotic membrane | Within 1-6 months after the start of the study
  intact or ruptured (accurate and wrong)
Fetal descent | Within 1-6 months after the start of the study
  -3,-2,-1,0,+1,+2,+3 (accurate and wrong)

CONTACTS AND LOCATIONS:
Overall Officials: Döndü BATKIN ERTÜRK, Principal Investigator — Midwifery
Locations (1):
- Tokat Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muliira RS, Seshan V, Ramasubramaniam S. Improving vaginal examinations performed by midwives. Sultan Qaboos Univ Med J. 2013 Aug;13(3):442-9. Epub 2013 Jun 25. PMID 23984031
- [Background] Chahine, E. B., Rizk, S., Young, M., Moynihan, A., Arluck, J., & Walker, P. (2018). Intern Bootcamp Cervical Dilation Simulation: Findings and Assessment [34M]. Obstetrics & Gynecology, 131, 150S.
- [Background] Pratinidhi, A., Patange, R., Patil, S., Salunkhe, J., & Samson, S. (2014). Testing of simulation training device for assessment of cervical dilatation among nursing student of Karad, India.
- [Background] https://www.internationalmidwives.org/assets/files/general-files/2019/10/icm-competencies-en-print-october-2019_final_18-oct-5db05248843e8.pdf erişim tarihi: 15.11.2019
- [Background] Arias T, Tran A, Breaud J, Fournier JP, Bongain A, Delotte J. A prospective study into the benefits of simulation training in teaching obstetric vaginal examination. Int J Gynaecol Obstet. 2016 Jun;133(3):380-4. doi: 10.1016/j.ijgo.2015.08.028. Epub 2016 Feb 23. PMID 26971257
- [Background] Cass GK, Crofts JF, Draycott TJ. The use of simulation to teach clinical skills in obstetrics. Semin Perinatol. 2011 Apr;35(2):68-73. doi: 10.1053/j.semperi.2011.01.005. PMID 21440813
- [Background] Bastable, S. B. (2017). Nurse as educator: Principles of teaching and learning for nursing practice. jones & bartlett learning
- [Background] Aslan, M. Günay, O. Çetinkaya, F. Mazıcıoğlu, M., (2002). Tıp Eğiticileri İçin Eğitim Becerileri Rehberi. Erciyes Üniversitesi Tıp Fakültesi, Yayın No:70, 80-88, Kayseri.
- [Background] McEwen BS, Sapolsky RM. Stress and cognitive function. Curr Opin Neurobiol. 1995 Apr;5(2):205-16. doi: 10.1016/0959-4388(95)80028-x. PMID 7620309
- [Background] Driscoll, Mp., (2005). Pyschology of Learning for İnstruction, 3rd Ed. New York: Pearson.
- [Background] Tiffen, J. Graf, N. Corbridge, S., (2009). Effectiveness of a Low-Fidelity Simulation Experience in Building Confidence Among Advanced Practice Nursing Graduate Students. Clinical Simulation in Nursing, 5(3), 113-117
- [Background] Nitsche JF, Shumard KM, Fino NF, Denney JM, Quinn KH, Bailey JC, Jijon R, Huang C, Kesty K, Whitecar PW, Grandis AS, Brost BC. Effectiveness of Labor Cervical Examination Simulation in Medical Student Education. Obstet Gynecol. 2015 Oct;126 Suppl 4:13S-20S. doi: 10.1097/AOG.0000000000001027. PMID 26375554
- [Background] Roosevelt L, Diebel M, Zielinski RE. Achieving competency in vaginal examinations: The challenge of balancing student learning needs with best practice in maternity care. Midwifery. 2018 Jun;61:39-41. doi: 10.1016/j.midw.2018.02.016. Epub 2018 Feb 23. PMID 29524775
- [Background] Abbas, A., Shaltout, A., & Fathalla, M. (2019). The Merit of Simulation in Teaching Medical Interns Vaginal Examination on Laboring Women. American Journal of Obstetrics And Gynecology, 220(1).